CLINICAL TRIAL: NCT04457544
Title: Spontaneous Coronary Artery Dissection (SCAD) National Swiss Registry (SwissSCAD)
Brief Title: Spontaneous Coronary Artery Dissection National Swiss Registry
Acronym: SwissSCAD
Status: Recruiting | Type: Observational
Sponsor: Dr. Sophie Degrauwe (Other)
Responsible Party: Sponsor-Investigator, Dr. Sophie Degrauwe, Doctor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2019-01886
Record Dates: First submitted 2020-06-16; First posted 2020-07-07 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Spontaneous Coronary Artery Dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective patients: The investigators will review the hospital records at the investigational site for SCAD events having occurred over the last 5 years. All SCAD patients aged ≥18 years, not presenting atherosclerotic or iatrogenic coronary dissection will be informed about the SwissSCAD study by phone and will be given at least one week to decide if they wish to participate. We plan to include 500 patients in the retrospective arm.
- Prospective patients: Patients presenting at the hospital with newly diagnosed SCAD will be informed of the SwissSCAD study and will be given at least one week to decide if they wish to participate. We plan to include 500 patients in the prospective arm.

SUMMARY:
Spontaneous coronary artery dissection (SCAD), is an underdiagnosed pathology, affecting predominantly young women without traditional cardiovascular risk factors and is associated with major adverse outcomes including myocardial infarction, cardiac arrest, or death.

Timely diagnosis of SCAD as well as clinical follow-up are of the essence in this pathology associated with major cardiac adverse outcomes. Despite recent improvements in diagnosis and recognition of the importance of SCAD, it remains poorly studied and understood.

In this context, we designed the SwissSCAD registry, a large, observational, prospective, cohort study, to describe the natural history of SCAD, its outcomes and its treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age.
* Patient presenting newly diagnosed SCAD or diagnosed with SCAD within the last 5 years.
* Subject must be willing to sign a Patient Informed Consent (PIC).

Exclusion Criteria:

* Patient unwilling or unable to provide informed consent.
* Patients with atherosclerotic or iatrogenic coronary dissection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This observational study will recruit consecutive male and female patients presenting with newly diagnosed SCAD or having been diagnosed with SCAD within the last 5 years.
  For the purposes of study inclusion, the definition of SCAD will be based on a central review of the coronary angiographic images confirmed by 2 independent assessors
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of safety events at 30 days | 30 days
  Incidence of Major cardiovascular outcomes (MACE) at 30 days

SECONDARY OUTCOMES:
Incidence of safety events at 1 year | 1 year
  Incidence of Major cardiovascular outcomes (MACE) at 1 year
Incidence of safety events at 5 years | 5 years
  Incidence of Major cardiovascular outcomes (MACE) at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Degrauwe, Dr, Principal Investigator — Hopitaux universitaires de Geneve
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided